CLINICAL TRIAL: NCT06359834
Title: Comparison of Remimazolam and Propofol Effect on Oxygen Reserve During Endoscopic Retrograde Cholangiopancreatography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4-2023-1693
Record Dates: First submitted 2024-04-07; First posted 2024-04-11 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Hepatobiiliary Diseases Requiring Endoscopic Retrograde Cholangiopancreatography
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam (Experimental): Patient group who receives remimazolam for sedation during endoscopy
  Interventions: Drug: Remimazolam besylate
- Propofol (Active Comparator): Patient group who receives propofol for sedation during endoscopy
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam besylate — Patients in this group receives 0.1mg/kg of remimazolam to induce sedation prior to endoscope insertion. Remimazolam 2mg is added in case of inadequate sedation.
  Arms: Remimazolam
Drug: Propofol — Patients in this group receives 1mg/kg of propofol to induce sedation prior to endoscope insertion. Propofol 20mg is added in case of inadequate sedation.
  Arms: Propofol

SUMMARY:
Propofol is one of the most commonly used sedative in endoscopic procedures, while its potency to induce respiratory depression may threaten patient safety. Remimazolam is known to less likely induce hemodynamic instability when compared to propofol, yet its favorable effects are not clearly evaluated in endoscopic procedures. Hence, this study aimed to compare hemodynamic effects of remimazolam and propofol, by evaluating oxygen reserve index (ORI) in patients scheduled for endoscopic retrograde cholangiopancreatography.

ELIGIBILITY:
Inclusion Criteria:

* Patients (age 19~80 yrs, ASA Class I~III) who are scheduled for elective endoscopic retrograde cholangiopancreatograph

Exclusion Criteria:

* Pregnancy Allergy to remimazolam or propofol Underlying pulmonary diseases or obstructive sleep apnea Underlying renal (serum Cr >2mg/dL) or cardiac disease (NYHA class III or IV) Hypotension (SBP <90mmHg) or hypoxemia (SpO2 <90%) assessed prior to procedure

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2024-04-11 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
Incidence of Oxygen Reserve Index (ORI) drop to 0.00 during sedation | Evaluation begins after sedative administration until the end of endoscopic procedure.
  Incidence of Oxygen Reserve Index (ORI) drop to 0.00 will be evaluated after sedative administration, until the end of endoscopic procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Gastroenterology, Department of Internal Medicine, Yonsei Institute of Gastroenterology, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim JH, Lee K, Lee SJ, Leem G, Lee HS, Park JY, Bang S, Park SW, Kim N, Chung MJ. Remimazolam Preserves Oxygen Reserve and Improves Sedation Safety Compared to Propofol in Endoscopic Retrograde Cholangiopancreatography. United European Gastroenterol J. 2025 Nov;13(9):1730-1739. doi: 10.1002/ueg2.70105. Epub 2025 Sep 5. PMID 40911638